CLINICAL TRIAL: NCT01924039
Title: Brief Motivational Enhancement Therapy for Individuals With Psychotic Disorders and Concurrent Substance Use Disorders
Brief Title: Brief Motivational Enhancement Therapy for Concurrent Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough study participants
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Yarissa Herman, Psychologist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 055/2013
Record Dates: First submitted 2013-08-07; First posted 2013-08-16 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Psychosis; Substance Use
Keywords: Psychosis; Substance Use; Motivational Enhancement Therapy
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Motivational Enhancement Therapy (Experimental)
  Interventions: Behavioral: Brief Motivational Enhancement Therapy
- treatment as usual (Other)
  Interventions: Behavioral: Brief Motivational Enhancement Therapy; Other: treatment as usual

INTERVENTIONS:
Behavioral: Brief Motivational Enhancement Therapy — The MET intervention consists of two 45 minute one-to-one sessions with a MET-trained therapist. The MET approach assists individuals to move through increasingly higher levels of change towards action (making change) and maintaining change. The MET approach aims to invoke rapid and internally motivated change with respect to substance use.
Other: treatment as usual — Treatment as usual includes case management as well as psychiatric appointments.
  Arms: treatment as usual

SUMMARY:
The investigators are proposing a project that will examine the effectiveness of brief motivational enhancement therapy in a population with concurrent psychotic disorders and substance use disorders. This study will represent an emerging line of inquiry, as best practice interventions with this concurrent disordered (CD) populations are yet to be established.

DETAILED DESCRIPTION:
Motivational enhancement therapy (MET) is grounded in research that explores the process of change. The MET approach assists individuals to move through increasingly higher levels of change towards action (making change) and maintaining change. The MET approach aims to invoke rapid and internally motivated change.

The Two MET sessions adapted from Sampl and Kadden (2001) are prepared as two individual sessions to reflect the original design of MET, allowing for client's to be met at their respective stage of change. Further, individual sessions allow the treatment to be tailored to client's individual reasons for change and personal coping strategies. The use of the Personalized Feedback Report (PFR) further encourages treatment around client's personal concerns and goals (Ramchand et al., 2011; See appendix 1 for further detail).

In the first treatment session, the therapist provides feedback from the initial CD consultation, using the PFR to stimulate discussion about personal substance use and reasons for change. Rapport building is also a key element to the first session, during which a strong therapeutic alliance is initiated. The second session is aimed at strengthening the commitment to change, exploring goal setting, and preparation for group.

The Centre for Addiction and Mental Health (CAMH) Schizophrenia Division introduced a CD service in 2009. Since the time of its inception, more than 200 consultations have been conducted. Of those consultations, more than 80%recommended attending CD groups offered with the Schizophrenia Program. However, less than 10% have followed those recommendations and attended the CD group.

Based on what is known about challenges surrounding engagement of CD clients in recommended treatments coupled with guidelines for evidence-based treatment with this population (Ledgerwood et al., 2008; Tsuang et al., 2006; Roncero et al., 2011), the purpose of the current study is to explore the ability of MET to increase engagement in CD interventions for clients diagnosed with psychotic and substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 16-65
* DSM-IV Diagnoses of a psychotic disorder and a substance use disorder (tobacco, alcohol and/or drug)
* Fluent English speaker
* Capable of giving written informed consent

Exclusion Criteria:

* Any medical or neuropsychiatric condition, illness or disorder (e.g. unstable angina, severe dementia) that could compromise attendance to outpatient appointments.
* Inability to provide informed consent.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
CD group attendance | 2 weeks
  The primary outcome engagement with outpatient CD service as measured by CD group attendance.

SECONDARY OUTCOMES:
Alcohol Use Scale (AUS)/Drug Use Scale (DUS) | 2 weeks and 3 months
  The secondary outcome is change in substance use as measured by the AUS and DUS

OTHER OUTCOMES:
Working Alliance Inventory | 2 weeks
  A measure of alliance between the participant and the clinician conducting the MET sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Yarissa Herman, D.Psych, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada